CLINICAL TRIAL: NCT06359496
Title: Split or Whole Liver Transplantation? A Multicenter Retrospective Cohort Study of Patients With Benign and Malignant Liver Disease
Status: Completed | Type: Observational
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Xiao Xu, Principal Investigator, Clinical Professor，PHD，MD, Zhejiang University
Other Study IDs: CT2024-ZJU-OBS8
Record Dates: First submitted 2024-04-04; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Zhejiang University
Keywords: liver transplantation; propensity score matching; split; whole; hepatocellular carcinoma; prognosis
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention factor — No intervention factor

SUMMARY:
The primary objective of this study was to assess the safety and feasibility of split liver transplantation(SLT) for adult hepatocellular carcinoma (HCC) patients, while comparing the prognostic disparities between adult SLT and WLT also .

Liver transplantation (LT) is an effective treatment for end-stage liver disease. As a traditional marginal donor liver, the application of SLT in pediatric patients is successful.However, its application in adult liver transplantation, especially in HCC patients, remains controversial.

This retrospective study analyze outcomes among adults who underwent SLT and whole liver transplantation (WLT) at two centers from January 2018 to August 2022. A 1:1 propensity score matching (PSM) analysis was performed based on important donor and recipient variables. Baseline characteristics and postoperative outcomes of the above recipients were analyzed and compared. Statistical significance was determined using a two-sided p-value threshold of less than 0.05.

DETAILED DESCRIPTION:
The primary objective of this study was to assess the safety and feasibility of split liver transplantation(SLT) for adult hepatocellular carcinoma (HCC) patients, while comparing the prognostic disparities between adult SLT and WLT also .

Liver transplantation (LT) is an effective treatment for end-stage liver disease. As a traditional marginal donor liver, the application of SLT in pediatric patients is successful.However, its application in adult liver transplantation, especially in HCC patients, remains controversial.

This retrospective study analyze outcomes among adults who underwent SLT and whole liver transplantation (WLT) at two centers from January 2018 to August 2022. A 1:1 propensity score matching (PSM) analysis was performed based on important donor and recipient variables. Baseline characteristics and postoperative outcomes of the above recipients were analyzed and compared. Statistical significance was determined using a two-sided p-value threshold of less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old
2. Received a liver transplantation between 2018 and 2022 (3) Liver transplantation was performed by SLT or WLT

Exclusion Criteria:

1. Re-LT
2. Multiorgan transplantation
3. Survival≤one week after LT
4. Incomplete data

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Each organ donation and transplantation strictly followed the guidelines of the Ethics Committee of the two hospitals, the current regulation of the Chinese Government and the Declaration of Helsinki. Every precaution has been taken to protect the privacy of research subjects and the confidentiality of their personal information. Informed consent was obtained from all patients.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2024-02-23 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-04-02 (Actual)

PRIMARY OUTCOMES:
Postoperative complications were evaluated by postoperative imaging reports and serological indicators | Jan.1 2018-Dec.31 2022
  Including rejection, emerging metabolic diseases, infections
The survival rate of each group was evaluated by follow-up survey and K-M curve | Jan.1 2018-Dec.31 2022
  Including overall survival rate and/or tumor free survival rate

CONTACTS AND LOCATIONS:
Locations (1):
- Xiao Xu, Hangzhou, China

IPD SHARING:
Plan to Share IPD: Yes
baseline characters of patients.
Supporting Information: SAP, CSR, Analytic Code
URL: http://www.cmm.zju.edu.cn/